CLINICAL TRIAL: NCT02037880
Title: Natural History Studies of Mucopolysaccharidosis III
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Sanfilippo Children's Research Foundation (Unknown); The Sanfilippo Research Foundation (Unknown); The Children's Medical Research Foundation (Unknown)
Responsible Party: Principal Investigator, Kevin Flanigan, MD, Nationwide Children's Hospital
Other Study IDs: MPSIII-1
Record Dates: First submitted 2013-11-26; First posted 2014-01-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Mucopolysaccharidosis Type IIIA; Mucopolysaccharidosis Type IIIB
Keywords: Mucopolysaccharidosis; MPS; Sanfilippo
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses | interventions — Spinal Puncture; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biobanking will include:
  1. Serum/Plasma
  2. Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MPS IIIA/B Subjects: Cohort will be followed for one year to assess natural history of the disease.
  Interventions: Procedure: Lumbar puncture; Device: Magnetic Resonance Imaging (MRI) of the brain

INTERVENTIONS:
Procedure: Lumbar puncture
Device: Magnetic Resonance Imaging (MRI) of the brain

SUMMARY:
The purpose of this study is to assess rates of decline in motor and cognitive functional measures, and to assess potential biomarkers, in order to identify potential outcome measure appropriate for use in therapeutic clinical trials.

DETAILED DESCRIPTION:
Mucopolysaccharidosis (MPS) type III (Sanfilippo syndrome) is a group of four devastating genetic diseases that result in the abnormal accumulation of glycosaminoglycans in body tissues. In MPSIII the predominant symptoms occur due to accumulation within the central nervous system (CNS), including the brain and spinal cord, resulting in cognitive decline, motor dysfunction, and eventual death.

In anticipation for future therapeutic studies for MPSIIIA and MPSIIIB, we are performing a natural history study to identify the following:

1. Individual rates of decline in motor and cognitive function in a cohort of potential clinical trial patients
2. The natural history of outcome measures in order to assess their appropriateness as outcomes in an eventual trial
3. Baseline functional data in patients who will be potential candidates for an eventual trial
4. Biomarkers of disease progression over a 12-month interval, including changes in brain MRI and in cerebrospinal fluid

Patients in this study will need to come to Nationwide Children's Hospital in Columbus, Ohio, three times. At each of these three time points, cognitive outcome measures will be assessed: at baseline (visit 1), 6 months (visit 2), and at 12 months (visit 3). At baseline (visit 1) and 12 months (visit 3), an MRI and a lumbar puncture will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 years old or greater
2. Confirmed diagnosis of MPSIIIA or MPSIIIB by either of two methods:

   1. No detectable or significantly reduced NAGLU (MPSIIIB) or SGSH (MPSIIIA) activity in serum or leukocyte assay
   2. Genomic DNA mutation analysis demonstrating a homozygous or compound heterozygous mutations in the NAGLU (MPSIIIB) or SGSH (MPSIIIA) genes
3. Clinical history of or examination features of neurologic dysfunction.

Exclusion Criteria:

1. Inability to participate in the clinical evaluations
2. Presence of a concomitant medical condition that precludes lumbar puncture or use of anesthetics
3. Inability to be safely sedated in the opinion of the clinical anesthesiologist

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals affected by MPS IIIA or MPS IIIB will be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cognitive function | up to 12 months
  Assessed using the Leiter International Performance assessment, a non-verbal assessment of cognitive function.

SECONDARY OUTCOMES:
Adaptive functioning | Months 0, 6, and 12
  Parental assessment of adaptive functioning using the Adaptive Behavioral Assessment System
Emotional/behavioral function | Months 0, 6, and 12
  Assessment of emotional/behavioral problems using the Child Behavioral Checklist
White and grey matter brain volumes | Months 0 and 12
  Assessment of brain volumes by MRI. MRI will be performed under sedation.

OTHER OUTCOMES:
Serum and cerebrospinal fluid NAGLU (MPSIIIB subjects) or SGSH (MPSIIIA subjects) levels | Months 0 and 12
  Measurement of NAGLU or SGSH activity in serum (by venipuncture) and CSF (by lumbar puncture). Lumbar puncture will be performed under sedation.
Liver size | Months 0 and 12
  Liver volume will be assessed by abdominal MRI obtained under the same sedation event as brain MRI and lumbar puncture.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Flanigan, MD, Principal Investigator — Nationwide Children's Hospital, Columbus, Ohio
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States